CLINICAL TRIAL: NCT05094479
Title: E-health Application in Supporting Lifestyle Changes During Pregnancy
Brief Title: E-health App and Lifestyle Changes During Pregnancy
Acronym: E-HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Business Finland (Other)
Responsible Party: Principal Investigator, Kirsi Laitinen, Associate Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-HEALTH
Record Dates: First submitted 2021-10-22; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Pregnancy; Dietary Habits; Physical Activity; Gestational Weight Gain
Keywords: Pregnancy; Health application; Diet quality; Physical activity; Gestational weight gain
MeSH Terms: conditions — Feeding Behavior; Motor Activity; Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health information delivered via health app (Experimental): Use of a health app with health information
  Interventions: Behavioral: Health information delivered via health app
- Control (No Intervention): Use of a health app without health information

INTERVENTIONS:
Behavioral: Health information delivered via health app — Intervention group will use a health app with non-personalized information on health-promoting lifestyle habits during pregnancy. Control group will use a health app without health information. Intervention effects on the lifestyle habits (gestational weight gain, diet quality, physical activity) will be investigated.
  Arms: Health information delivered via health app

SUMMARY:
The purpose of this online follow-up study is to investigate health app use in pregnant women and through a pilot intervention trial investigate whether the addition of evidence-based information on health-promoting lifestyle delivered via the health app has an effect on lifestyle habits (gestational weight, diet quality and physical activity) during pregnancy.

DETAILED DESCRIPTION:
An online follow-up study with a 2-arm equal allocation parallel randomized controlled pilot intervention trial with pregnant women (n=1000) will be conducted. The intervention consists of non-personalized, evidence-based information on health-promoting lifestyle during pregnancy delivered via a health app. Control group uses the health app without health information.

Aims of an exploratory part of the study are to characterize the health app use and users among pregnant women and to investigate whether the frequency of the health app use during pregnancy has an effect on lifestyle habits. Aim of the pilot intervention is to investigate whether the addition of evidence-based information on health-promoting lifestyle delivered via the health app has an effect on lifestyle habits during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, less than 28 pregnancy weeks
* Fluency in Finnish

Exclusion Criteria:

* Not pregnant
* No fluency in Finnish

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females
Enrollment: 1047 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Change in gestational weight | Pre-pregnancy weight reported at enrollment and current weight at late pregnancy (pregnancy weeks 35-36)
  Self-reported weight assessed by a questionnaire
Change in diet quality scores | At enrollment and late pregnancy (pregnancy weeks 35-36)
  Assessed by a validated Index of Diet Quality (IDQ); scores range from 0 to 15 points with higher scores meaning better diet quality.

SECONDARY OUTCOMES:
Change in physical activity scores | At enrollment and late pregnancy (pregnancy weeks 35-36)
  Assessed by a validated metabolic equivalent (MET)-index; scores range from 0 to 105 MET h/wk with higher scores meaning more vigorous physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi Laitinen, Assoc. Prof., Principal Investigator — University of Turku
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No